CLINICAL TRIAL: NCT02854202
Title: Effect of High Protein Breakfast on Overall Postprandial Glycemia in Type 2 Diabetes
Brief Title: High Protein Breakfast on Postprandial Glycemia in T2D (PBD)
Acronym: PBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas Caracas (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, MD, Professor, Hospital de Clinicas Caracas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCBI 017-2008-112
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1-Whey protein (Experimental): In the Arm 1-Whey protein Breakfast the participant will consume 42 g protein at breakfast mainly from whey
  Interventions: Other: Arm1: Whey protein
- Arm 2 Breakfast- other proteins (Active Comparator): In the Arm 2 Breakfast- other proteins sources (No Whey) the participants will consume 42 g protein from other sources (no Whey) at breakfast
  Interventions: Other: Arm 2 Breakfast- other proteins
- Arm 3 Breakfast- low protein (Placebo Comparator): In the Arm 3: breakfast with low proteins content, the participant will consume 22 g protein at breakfast
  Interventions: Other: Arm 3 Breakfast- low protein

INTERVENTIONS:
Other: Arm1: Whey protein — Arm1: Whey protein:The participants will consume 42 g protein, namely from Whey protein in the breakfast
  Other Names: WB
  Arms: Arm 1-Whey protein
Other: Arm 2 Breakfast- other proteins — Arm 2 Breakfast- other proteins: The participants will be assigned to 42 g protein of other protein sources at breakfast
  Other Names: PB
  Arms: Arm 2 Breakfast- other proteins
Other: Arm 3 Breakfast- low protein — Arm 3: Low protein' :The participants will consume 22 g protein at breakfast
  Other Names: LP
  Arms: Arm 3 Breakfast- low protein

SUMMARY:
The investigators hypothesis is that eating whey protein in breakfast will reduce overall postprandial glycemia in individuals with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
It was shown that increasing protein at breakfast results in reduced overall postprandial glycemia in obese individuals This study was undertaken to evaluate whether compared to proteins like tuna, eggs and soy, the intake of whey protein in the breakfast is more effective to reduce overall postprandial glycemia (PPHG) in T2D individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Participants: from 30 to 72 years of age
2. BMI: 26 to 34 kg/m2)
3. Diabetes criteria
4. HbA1C: 7-9 % or
5. Habitually eat breakfast
6. Only naïve or treated with metformin.
7. Not dieting and no change in body weight >10 lb = 4.5 kg within the last 3 months
8. Normal liver, kidney and thyroid function.

Exclusion Criteria:

1. Type 1 Diabetes
2. Anemia (Hg > 10 g/dL)
3. Serum creatinine level < 1.5 mg/dl
4. Pulmonary disease, psychiatric, immunological, neoplastic diseases or severe diabetic complications, such as cardiovascular disease, cerebrovascular disease, proliferative diabetic retinopathy, gastroparesis or underwent bariatric surgery.
5. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase and/or aspartate
6. Infectious disease
7. Pregnant women or lactating
8. Known hypersensitivity to milk components
9. Documented or suspected history (within one year) of illicit drug abuse or alcoholism.

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | 3 month
  Overall postprandial glycemia after breakfast, lunch and dinner

SECONDARY OUTCOMES:
Satiety | 3 month
  Postprandial satiety after breakfast lunch and dinner, assessed with visual analog scale.
Change in body weight | 3 month
  Body weight will be assessed every every two weeks during 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Wolfson Medical Center

IPD SHARING:
Plan to Share IPD: No